CLINICAL TRIAL: NCT01630720
Title: Vitamin Therapy in JGH Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, John Hoffer, MD, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-041
Record Dates: First submitted 2011-06-21; First posted 2012-06-28 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Patients With Hypovitaminosis C and D; Vitamin Deficiencies
Keywords: ascorbic acid; cholecalciferol; vitamin C; vitamin D; hypovitaminosis; mood; distress
MeSH Terms: conditions — Avitaminosis | interventions — Ascorbic Acid; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin C (Active Comparator): vitamin C 500 mg twice daily
  Interventions: Dietary Supplement: vitamin C or vitamin D
- vitamin D (Active Comparator): vitamin D 5000 IU daily
  Interventions: Dietary Supplement: vitamin C or vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin C or vitamin D — vitamin C 500 mg twice daily versus vitamin D 5000 IU daily for 7 to 10 days

SUMMARY:
There is a high prevalence of hypovitaminosis C and D in our hospital and other acute-care hospitals. Since the correction of these presumed deficiency states is simple, safe and inexpensive, their documented or suspected presence would normally be considered sufficient indication to correct them. However, the common practice is to ignore them. Identification of specific measurable medical consequences of hypovitaminosis C or D would provide a stronger case to treat or prevent in-hospital vitamin deficiency states.

Biochemical deficiencies of vitamin C and D have both been linked to mood disturbance, and hypovitaminosis C reportedly increases blood histamine concentrations.

We recently found that the provision of vitamin C (500 mg twice daily) but not vitamin D (1000 IU twice daily) promptly improved the average mood score of acutely hospitalized patients. We will now conduct a closely similar randomized clinical trial using a more adequate dose of vitamin D, namely 5000 IU/day for up to 10 days.

DETAILED DESCRIPTION:
HYPOTHESIS:

Adequate vitamin C or vitamin D provision to mentally competent acutely hospitalized patients for 7 to 10 days will correct their biochemical deficiency, improve their mood, and (in the vitamin C-treated patients) reduce blood histamine concentrations.

PROTOCOL:

1. Mentally competent patients fluent in English or French admitted to the surgical or medical units of the hospital will be offered participation.
2. Plasma vitamin C and 25-hydroxyvitamin D, serum C-reactive protein, parathyroid hormone level (a measure of vitamin D adequacy) and blood histamine will be measured in participating patients prior to starting the treatment and after 7 to 10 days of treatment.
3. Within 24 h prior to and within 24 after the 5-10 d treatment course the patient will complete the POMS-B, a validated one-page 30-item questionnaire that assesses mood and energy, and the Distress Thermometer. Patients followed only for the 5-10 d duration of the clinical trial.
4. The chart will be reviewed for age, sex, diagnosis, and pertinent lab results.
5. After the initial blood sample has been drawn and the questionnaire completed the patient will begin treatment either with vitamin C 500 mg twice daily or vitamin D 5000 IU daily; both vitamins will be prescribed by one of the collaborating physicians without knowledge of the person who recruits, assesses and follows the patient. Treatment assignment will be by coin toss.

7. The questionnaire and blood sampling will be repeated after 7 to 10 days of treatment (as determined by feasibility and the situation on the ward) or prior to discharge if discharge is going to occur before the full course of treatment.

8. Neither the patient nor the person who administers the questionnaires will know which patient receives vitamin C or D. The vitamin D and C tablets are distinguishable, so patients motivated to do so could figure out which vitamin they are being prescribed. Since both treatments are being used to correct deficiency diseases which are strongly suspected to affect mood, neither patients, nurses, nor the students following the patients have no basis to anticipate that one treatment will improve their mood more than the other one.

ELIGIBILITY:
Inclusion Criteria:

* acutely hospitalized in our hospital
* mentally competent
* judged likely to remain in hospital for at least the following 7 days
* fluent in French or English

Exclusion Criteria:

* presence of hypercalcemia
* receiving hemodialysis treatment
* critically ill
* unable to take medication by mouth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
mood | prior to and after 5-10 days of treatment
  total mood disturbance score on the POMS-B (profile of mood states). Durations of hospital stay are variable and often unpredictable. The intended duration of therapy is 7 to 10 days of treatment, with baseline just prior to starting and outcome measurement recorded just after the final day of therapy. The 7-10 day window is necessary and valid to account for vagaries in duration of hospital stay as well as the interfering effect of weekends when less staffing is available. As in our prior published work, any treatment duration 5 days or longer is included as sufficient.

SECONDARY OUTCOMES:
Blood histamine concentration | prior to and after 5-10 days of treatment
  Blood histamine concentration. Durations of hospital stay are variable and often unpredictable. The intended duration of therapy is 7 to 10 days of treatment, with baseline just prior to starting and outcome measurement recorded just after the final day of therapy. The 7-10 day window is necessary and valid to account for vagaries in duration of hospital stay as well as the interfering effect of weekends when less staffing is available. As in our prior published work, any treatment duration 5 days or longer is included as sufficient.
distress | prior to and after 5-10 days of treatment
  the distress thermometer. Durations of hospital stay are variable and often unpredictable. The intended duration of therapy is 7 to 10 days of treatment, with baseline just prior to starting and outcome measurement recorded just after the final day of therapy. The 7-10 day window is necessary and valid to account for vagaries in duration of hospital stay as well as the interfering effect of weekends when less staffing is available. As in our prior published work, any treatment duration 5 days or longer is included as sufficient.

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Wang Y, Liu XJ, Robitaille L, Eintracht S, MacNamara E, Hoffer LJ. Effects of vitamin C and vitamin D administration on mood and distress in acutely hospitalized patients. Am J Clin Nutr. 2013 Sep;98(3):705-11. doi: 10.3945/ajcn.112.056366. Epub 2013 Jul 24. PMID 23885048